CLINICAL TRIAL: NCT04013802
Title: Administration of Most Closely HLA-matched Multivirus-specific Cytotoxic T-Lymphocytes for the Treatment of EBV, CMV, Adenovirus, and BK Virus Infections Post Allogeneic Stem Cell Transplant
Brief Title: TETRAVI Multivirus CTL for Treatment of EBV, CMV, Adenovirus, and BK Infections Post Allogeneic SCT.
Acronym: TETRAVI
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, John Craddock, Associate Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-44843 TETRAVI
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Viral Infection
Keywords: cytomegalovirus (CMV); BK virus; Epstein-Barr virus (EBV); adenovirus
MeSH Terms: conditions — Virus Diseases; Epstein-Barr Virus Infections; Adenoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- HLA-matched VSTs (Experimental): Partially HLA-matched VSTs will be thawed and given by intravenous injection. Patients will receive 2 x 10^7 or 4 x 10^7 partially HLA-matched MVSTs, depending on their body surface area, as a single infusion. In the rare case where insufficient banked cell product is available, a lower number of cells may be infused with agreement of the principal investigator, patient and/or guardian and the treatment team
  Additional doses may be from the same donor or a different donor based on available cell lines and patient/disease factors. Decision to switch to a different donor can be made by the principal investigator based on factors that include sequential treatment of different viral infections, concerns for immune escape of the targeted virus and/or availability of a better matched or otherwise superior VST line. Additional treatments will only be given following the agreement of the patient, treating physician, and investigator. This process can be repeated as needed.
  Interventions: Biological: HLA-matched VSTs

INTERVENTIONS:
Biological: HLA-matched VSTs — An alternative approach that bypasses the need to grow VSTs for individual patients is to bank closely HLA-matched allogeneic VSTs that could be available as an "off the shelf" product.
  The HLA-matched VST product is to produce immune activity to CMV, Adv, BK virus and EBV in all recipients.
  Most recently our group extended this "off the shelf" approach to five viruses using the T cell product manufactured in 10 days. The VSTs were administered to 38 patients with 45 infections in a phase II clinical trial. A single infusion produced a cumulative complete or partial response rate of 92% overall and the following rates by virus: 100% for BKV (n = 16), 94% for CMV (n = 17), 71% for AdV (n = 7), 100% for EBV (n = 2), and 67% for HHV-6 (human herpesvirus) (n = 3).

SUMMARY:
The purpose of this study is to use VSTs (virus-specific T cells) from a donor that is a partial HLA (human leukocyte antigen) match with the patient to treat viral infections after an allogeneic hematopoietic stem cell transplant (HSCT). These cells may also have value in CAR-T recipients who have received a product that depletes virus specific T cells.

The patient must have had a myeloablative or non-myeloablative allogeneic HSCT using either bone marrow, single/double umbilical cord blood, or peripheral blood stem cells (PBSC) or CAR T cell product targeting an antigen expressed on virus specific T cells. After a transplant, while the immune system grows back, the patient is at risk for infection. Some viruses can stay in the body for life and are normally controlled by a healthy immune system, but if the immune system is weakened, like after a transplant, they can cause life threatening infections. He/she must have had an infection with one or more of the following viruses -Epstein Barr virus (EBV), cytomegalovirus (CMV), adenovirus (AdV), Human polyomavirus type I (BKV), and human polyomavirus type II (JCV)- that has persisted or recurred despite standard therapy.

In this study, the investigators want to use white blood cells that have been trained to treat viral infections. In an earlier study the investigators showed that treatment with such specially trained T cells has been successful when the cells are made from the transplant donor. However as it takes 1-2 months to make the cells, that approach is not practical for patients who already have an infection. In a subsequent study, the investigators were able to create multivirus-specific T cells (VSTs) from the blood of healthy donors and created a bank of these cells. The investigators then successfully used these banked cells to treat virus infections after a stem cell transplant. In this study the investigators have further modified their production method to decrease the potential side effects and the investigators want to find out if they can use these banked VSTs to fight infections caused by the viruses mentioned above.

DETAILED DESCRIPTION:
The virus-specific T cells (VSTs) given to the patient will be thawed and injected into their intravenous line. To prevent an allergic reaction if the patient had a prior reaction to blood products like blood transfusions or platelets, prior to receiving the VSTs he/she may be given diphenhydramine (Benadryl) and acetaminophen (Tylenol). The patient will remain in the clinic for at least one hour after the infusion.

If the patient has persistent infection after the first dose, the investigators would discuss this with the patient and allow them to receive additional treatments if there were no complications with prior infusions. These additional treatments might be with cells from the same donor, or if the investigators feel that there is another donor whose cells might be better for the patient, the investigators would use cells from a different donor. This second product will be administered at the same dose level 14 days after the patient's initial infusion, and any additional infusions should be at least 14 days apart. After each VST infusion, the patient will be monitored as described above.

After the patient receives the cells the patient's transplant doctor will monitor the levels of the virus the subject is infected with in their blood.

The patient will continue to be followed by their doctor(s) after the injection. They will be seen in the clinic by research staff for follow up every week for 6 weeks. To learn more about the way the VSTs are working in the patient's body, up to an extra 30-40 ml (6-8 teaspoons) of blood may be taken before the infusion and at week 1 (optional), 2, 4, and 6. Blood should come from the central intravenous line, and should not require extra needle sticks. Depending on clinical and laboratory response, samples may be collected at additional time points.

Any leftover samples of blood may be used to help future research. The specimens may be kept for a long time. These specimens and information about the patient's circumstances may be shared with other cancer researchers. Although there will be a record identifying under what circumstances these specimens were obtained, under all circumstances the patient's identity will be kept confidential.

Study Duration: The patient will be on the study for approximately one year after their VST infusion. If the patient receives additional doses of the T cells as described above, the patient will be followed for one year after their last dose of T-cells.

ELIGIBILITY:
Inclusion Criteria:

1. Prior myeloablative or non-myeloablative allogeneic hematopoietic stem cell transplant using either bone marrow or peripheral blood stem cells or single or double cord blood.

   Or Received CAR-T cells targeting an antigen expressed on normal virus specific T cells
2. Treatment for Infection/Disease will fall into one of 3 categories (options):

   * Option 1: Persistent, increasing or recurrent infections despite 7 days of standard therapy;

     * a. CMV: Treatment of persistent or relapsed CMV disease or infection after standard therapy. For CMV infection, standard therapy is defined as antiviral therapy with ganciclovir, foscarnet, letermovir or cidofovir. 56, 57

       * i. CMV disease: defined as the demonstration of CMV by biopsy specimen from visceral sites (by culture or histology) or the detection of CMV by culture or direct fluorescent antibody stain in broncheoalveolar lavage fluid in the presence of new or changing pulmonary infiltrates or changes consistent with CMV retinitis on ophthalmologic examination.
       * ii. CMV infection: defined as the presence of CMV positivity as detected by PCR or pp65 antigenemia or culture from ONE site such as stool or blood or urine or nasopharynx or bronchoalveolar lavage.
     * b. Adenovirus: Treatment of persistent adenovirus infection or disease despite standard therapy. Standard therapy is defined as antiviral therapy with cidofovir.

       * i. Adenovirus infection: defined as the presence of adenoviral positivity as detected by PCR or culture from ONE site such as stool or blood or urine or lung or nasopharynx.
       * ii. Adenovirus disease: defined as the presence of adenoviral positivity as detected by PCR, DFA or culture from two or more sites such as stool or blood or urine or lung or nasopharynx.
     * c. EBV: For treatment of persistent EBV infection despite standard therapy. For EBV infection, standard therapy is defined as rituximab given at 375mg/m2 in patients for 1-4 doses with a CD20+ve tumor.58

       * i. EBV infection: defined as: (1) Biopsy proven lymphoma with EBV genomes detected in tumor cells by immunocytochemistry or in situ PCR;
       * ii. (2) Or clinical or imaging findings consistent with EBV lymphoma and/or elevated EBV viral load in peripheral blood.
     * d. BK virus: Treatment of persistent BK virus infection or BK virus disease despite antiviral treatment with cidofovir or leflunomide. No clear standard treatment is defined (section 1.1.5). Cidofovir has been administered in low doses as well as high doses to HSCT patients with BK infections but no randomized trials are available proving its clinical efficacy.

       * i. BK virus infection is defined as the presence of BK virus positivity as detected by PCR or culture in one site such as blood or urine or lung.
       * ii. BK virus disease is defined as the presence of BK virus detectable by culture or PCR in blood or urine or other body fluids or lungs and symptoms of disease including, but not limited to persistent microscopic or macroscopic hematuria or detectable BK virus in more than one site.
     * e. JC virus: Treatment of JC virus infection or disease without suitable alternative treatment option. Given the high homology (>90%) between JC and BK and the fact that BKVSTs targeting VP1 and Large T (as targeted in our multivirus MVSTs) have been administered to treat JCV-PML, and produced viral clearance from the cerebrospinal fluid, it is likely that our MVSTs will have efficacy against JC virus. Given the current lack of treatment options for JC virus infection or reactivation after HSCT and the risk of progression to JML, which is almost uniformly fatal, and the apparent activity of BK virus- directed T cells against JC virus infected cells, we propose including patients with JC virus on this study, unless a suitable alternative therapy is available.

       * i. JC virus infection is defined as the presence of elevated JC virus levels as detected by PCR or positive culture in one site such as CSF or blood.
       * ii. JC virus disease is defined as defined as the presence of JC virus detectable by culture or PCR in one or more sites such as blood or CSF and symptoms of disease including symptoms of PML OR detectable JC virus by PCR or culture in more than one site.
   * Option 2: Early treatment for single or multiple infections with EBV, CMV, adenovirus, and/or BK virus will be allowed for patients deemed to be unable to tolerate standard therapy. Patients with multiple CMV, EBV, Adenovirus, and BK virus infections are eligible given that at least one infection is persistent despite standard therapy as defined above. Patients with multiple infections or reactivations are eligible to enroll.
   * Option 3: For patients having adenovirus and BK virus, the requirement to fail one week of standard therapy would be waived if they meet one of the criteria below:

     1. They are ≤100 days post- transplant
     2. They are currently receiving other nephrotoxic agents or marrow-suppressive agents
     3. They have adenovirus copy number ≥10,000 copies/ml
3. Clinical status at enrollment to allow tapering of steroids to equal or less than 0.5 mg/kg/day methylprednisolone (or equivalent).
4. Hgb ≥ 7.0 gm/dl
5. Available MVSTs must be partially HLA matched with recipient and HLA match must be verified by one of the Principal Investigators.
6. Negative pregnancy test in female patients if applicable (childbearing potential who have received a reduced intensity conditioning regimen).
7. Written informed consent and/or signed assent line from patient, parent or guardian.

Exclusion Criteria

1. Patients receiving ATG, Campath or other immunosuppressive T cell monoclonal antibodies within 28 days of screening for enrollment.
2. Patients with other uncontrolled infections. For bacterial infections, patients must be receiving definitive therapy and have no signs of progressing infection for 72 hours prior to enrollment. For fungal infections patients must be receiving definitive systemic anti-fungal therapy and have no signs of progressing infection for 1 week prior to enrollment.

   Progressing infection is defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.
3. Patients who are less than 28 days removed from their allogeneic hematopoietic stem cell transplant or who have received donor lymphocyte infusions (DLI) or CAR-T within 28 days.
4. Patients with active acute GVHD grades II-IV.
5. Uncontrolled relapse of malignancy
6. Requirement for FiO2 > 50% oxygen to maintain oxygen saturation > 90% (peripheral pulse-ox). Note: patients requiring oxygen at FiO2<=50% to maintain arterial oxygen saturation >90% are eligible to receive MVSTs if the reason for this oxygen requirement is believed attributable to the virus being treated.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2031-05-01 (Estimated)

PRIMARY OUTCOMES:
Treatment related adverse events. | 28 days after the last dose of MVST
  The primary objective is to measure the safety of MVSTs based on patients with grades 3-5 non-hematologic adverse events that are at least possibly related to the T cell product.

SECONDARY OUTCOMES:
Number of patients with acute GvHD. | 42 days after the last dose of MVST
  Patients with acute GvHD grades III-IV, summarized by the proportion of patients with acute GvHD grades III-IV among all safety evaluable patients.
Antiviral Response. | 42 days following the last treatment of MVST
  The antiviral response is defined as the viral load reduction by at least 50% (partial response) or return to the normal level (complete response) for the treated virus (at least one of the 4 virus types: CMV, EBV, adenovirus, and BK virus). The antiviral response rate is defined as the proportion of subjects with a partial or complete response among all response evaluable patients.
Number of patients with secondary graft failure. | 42 days following the last treatment of MVST
  Secondary graft failure is defined as initial neutrophil engraftment followed by subsequent decline in the ANC to less than 500/mm3 for three consecutive measurements on different days, unresponsive to growth factor therapy and persists for at least 14 days in the absence of a known cause such as relapse.

CONTACTS AND LOCATIONS:
Overall Officials: John Craddock, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No